CLINICAL TRIAL: NCT06415890
Title: The Effect of Usıng The 4-7-8 Breathıng Technıque on Postoperatıve Shoulder Paın and Respıratory Functıon Tests After Laparoscopıc Cholecystectomy
Brief Title: Effect of 4-7-8 Breathıng Technıque on Shoulder Paın and Respıratory Functıon Tests After Laparoscopıc Cholesectectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Ayse Nur Serbest Baz, Lecturer, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HMKU-SERBEST-001
Record Dates: First submitted 2024-05-05; First posted 2024-05-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Laparoscopic Cholecystectomy; Breathing Exercise; Pulmonary Function Test; Shoulder Pain; Surgical Nursing; 4-7-8 Breathing Technique
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-arm randomized controlled clinical trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The information that the patients included in the research sample were assigned to groups A and B according to the randomization table will be kept by the consultant, the researcher will fill out the "Informed Consent Form" for all patients when he/she goes to the patient for the application, and then the consultant will share the information about which group the patient is in with the researcher. When the research is completed, the data will be transferred to the computer environment by a statistician who does not know the A and B groups and the data will be analyzed by a statistician independent of the research and the findings will be reported. Thus, the data analysis and statistics phase will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercise Group (Experimental): In addition to the routine treatment and care practices of the clinic, the patients included in the study group will be taught the 4-7-8 breathing technique by the researcher and applied after surgery. They will be provided to complete one set (4 breaths) by practicing the 4-7-8 breathing technique first with the researcher and then alone. The training will last approximately 15 minutes for each patient. Patients will be asked to start the first breathing exercise at the 4th hour after coming to the clinic after laparoscopic cholecystectomy and perform one set (4 breaths) every two hours.
  Interventions: Other: 4-7-8 Breathing Technique
- Control Group (No Intervention): Patients in the control group will receive routine treatment and care after laparoscopic cholecystectomy. In the clinic, patients are not trained on postoperative breathing exercises and the use of triflow is recommended. However, there is no planned training for the use of this tool and the patients' use of the tool is not monitored.

INTERVENTIONS:
Other: 4-7-8 Breathing Technique — The 4-7-8 breathing technique to be applied to the patients in the experimental group; the patient will be asked to sit or lie in a comfortable position with his/her hands on his/her lap, press the tip of his/her tongue on the tissue protrusion behind the upper front teeth and hold it there during the breathing cycle, breathe in through the nose for four counts, hold the breath for seven counts and then slowly exhale through the mouth for eight counts and complete a set. Within one set of practice, this cycle repeats four times.
  Arms: Breathing Exercise Group

SUMMARY:
This study was planned as a randomized controlled clinical trial to determine the effect of 4-7-8 breathing technique on shoulder pain and pulmonary function tests after laporoscopic cholecystectomy. A sample of 96 patients will be randomly assigned to the study and control groups. The study group will be administered the 4-7-8 breathing technique after LK, while the control group will be given routine care of the ward. Shoulder pain and pulmonary function tests will be measured in the first 24 hours and at discharge. The data obtained will be analyzed by appropriate statistical methods.

DETAILED DESCRIPTION:
Laporoscopic cholecystectomy (LC) is the most commonly used method for the treatment of cholecystitis, one of the most common diseases of the digestive system. In addition to its advantages such as low risk of complications and usually requiring less than 24 hours of hospitalization, shoulder pain develops in approximately 35-80% of patients after LC. After LK, patients' lungs may be affected due to factors such as intraoperative general anesthesia, mechanical ventilation support, carbon dioxide (CO2) pneumoperitoneum administration, anesthetic drugs and patient positioning, and patients experience shoulder pain, especially with CO2 pneumoperitoneum administration. In patients undergoing LK, shoulder pain felt throughout the thorax causes spasm and restriction of movement in the muscles assisting respiration and an increase in intercostal tone. This leads to a decrease in the amount of air filling the lungs, accumulation of secretions, pneumonia, decreased functional residual volume and increased risk of atelectasis. For this reason, it is necessary to evaluate the respiratory system in patients undergoing LK as in all surgical interventions and to monitor pulmonary functions (FVC, FEV1, FEV1/FCV) to evaluate the deterioration in lung functions and to control pain with pharmacologic and non-pharmacologic methods. One of the respiratory exercises that nurses can apply independently in the removal of CO₂, improvement of respiratory functions and pain control after surgery is the 4-7-8 breathing technique. This technique has been proven to have positive contributions in pain control, and its easy application, reliability and non-invasiveness make its use widespread.

This study was planned as a randomized controlled clinical trial to determine the effect of 4-7-8 breathing technique on shoulder pain and pulmonary function tests after LK. A sample of 96 patients will be randomly assigned to the study and control groups. The study group will be administered the 4-7-8 breathing technique after LK, while the control group will be given routine care of the ward. Shoulder pain and pulmonary function tests will be measured in the first 24 hours and at discharge. The data obtained will be analyzed by appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective laparoscopic cholecystectomy,
* Admitted to the clinic at least 2 hours before the surgical procedure,
* Open to communication and cooperation,
* Written and verbal permission to participate in the study was obtained,
* Conscious, oriented and cooperative,
* No cognitive and mental problems,
* Speaks and understands Turkish,
* American Society of Anesthesiologists (ASA) classification scores of I and II,
* Hospitalized at least one night after surgical intervention,
* Patients aged 18 years and older will be included in the study.

Exclusion Criteria:

* Undergoing emergency laparoscopic cholecystectomy,
* Open cholecystectomy,
* Not admitted to the clinic at least 2 hours before the surgical procedure,
* Not open to communication and cooperation,
* Written and verbal permission to participate in the research could not be obtained,
* Unconscious, disoriented and uncooperative,
* Cognitively and mentally impaired,
* Speaking Turkish but not understanding it,
* Discharged on the same day after surgical intervention,
* ASA score III and above,
* Patients aged 18 years and younger will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain | Second postoperative day
  Visual Analog Scale (VAS):The VAS used in this study is a one-dimensional pain scale commonly used in adult populations. The VAS is a continuous scale consisting of a horizontal or vertical line 10 centimeters (100 mm) long. Pain intensity is determined by statements ranging from "no pain" at one end of the scale to "excruciating pain" at the other end. The participant is asked to place a line perpendicular to the VAS line at the point representing pain intensity. Pain scoring is determined by measuring the distance (mm) on the 10-centimeter line using a ruler and is defined by providing a score range between 0-100 mm (No pain=0-4 mm, mild pain=5-44 mm, moderate pain=45-74 mm and severe pain=75-100 mm). In this study, the vertical form of the VAS will be used to evaluate shoulder pain in patients after surgical intervention based on the information that the vertical form of the VAS gives more accurate results than the horizontal form
  Translated with DeepL.com (free version)
Pulmonary Function Test | Second postoperative day
  Pulmonary Function Test: Pulmonary function values will be evaluated with a portable . FVC (%), FEV1 (%) and FEV1/FVC (%) parameters will be used in the evaluationpulmonary function test device.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay ALTUN UĞRAŞ, Study Director — Mersin University
Locations (1):
- İskenderun Devlet Hastanesi, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hosseinzadeh F, Nasiri E, Behroozi T. Investigating the effects of drainage by hemovac drain on shoulder pain after female laparoscopic surgery and comparison with deep breathing technique: a randomized clinical trial study. Surg Endosc. 2020 Dec;34(12):5439-5446. doi: 10.1007/s00464-019-07339-z. Epub 2020 Jan 13. PMID 31932939
- [Background] Aktas GK, Ilgin VE. The Effect of Deep Breathing Exercise and 4-7-8 Breathing Techniques Applied to Patients After Bariatric Surgery on Anxiety and Quality of Life. Obes Surg. 2023 Mar;33(3):920-929. doi: 10.1007/s11695-022-06405-1. Epub 2022 Dec 8. PMID 36480101
- [Background] Chinagudi, S., Badami, S., Herur, A., Patil, S., Gv, S., & Ankad, R. (2014). Immediate effect of short duration of slow deep breath-ing on heart rate variability in healthy adults. National Journal of Physiology, Pharmacy and Pharmacology, 4(3), 233- 235.
- [Background] Vierra J, Boonla O, Prasertsri P. Effects of sleep deprivation and 4-7-8 breathing control on heart rate variability, blood pressure, blood glucose, and endothelial function in healthy young adults. Physiol Rep. 2022 Jul;10(13):e15389. doi: 10.14814/phy2.15389. PMID 35822447
- [Background] Toleska M, Dimitrovski A, Shosholcheva M, Kartalov A, Kuzmanovska B, Dimitrovska NT. Pain and Multimodal Analgesia in Laparoscopic Cholecystectomy. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2022 Jul 13;43(2):41-49. doi: 10.2478/prilozi-2022-0017. PMID 35843915
- [Background] Lee J, Hur MH. The Effects of Aroma Essential Oil Inhalation on Stress, Pain, and Sleep Quality in Laparoscopic Cholecystectomy Patients: A Randomized Controlled Trial. Asian Nurs Res (Korean Soc Nurs Sci). 2022 Feb;16(1):1-8. doi: 10.1016/j.anr.2021.11.002. Epub 2021 Dec 24. PMID 34954406
- [Background] Russo MA, Santarelli DM, O'Rourke D. The physiological effects of slow breathing in the healthy human. Breathe (Sheff). 2017 Dec;13(4):298-309. doi: 10.1183/20734735.009817. PMID 29209423